CLINICAL TRIAL: NCT06841497
Title: Safety and Efficacy Assessment of Unani Formulation 'Dolabi' in Management of Diabetes Mellitus Type II
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hamdard University (Other)
Responsible Party: Principal Investigator, Abdul Bari, Principal Investigator, Hamdard University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DLB-PII-HLWP
Record Dates: First submitted 2025-02-17; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Diabetes Mellitus; Type 2 DM
Keywords: Diabetes Mellitus; T2DM; Metabolic disease; Insulin Resistance
MeSH Terms: conditions — Diabetes Mellitus; Metabolic Diseases; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Effect of Dolabi on DM II (Experimental)
  Interventions: Other: Dolabi

INTERVENTIONS:
Other: Dolabi — herbal remedy for DM II

SUMMARY:
Diabetes is a chronic health condition that affects millions of people worldwide. In recent years, Pakistan has witnessed a significant increase in the prevalence of diabetes, making it a major public health concern. To address this growing problem, conducting clinical trials on diabetes in Pakistan is of utmost importance. Clinical trials play a crucial role in advancing medical knowledge, improving patient care, and finding effective treatments for diabetes.

This research aims to assess the safety and effectiveness of the Unani formulation Dolabi in treating type II diabetes mellitus. The study consists of two phases: a pre-clinical phase, which involves acute and subacute oral toxicity testing on animal models, and a clinical phase, which includes a single-blind, single-arm, multicenter, phase II clinical trial conducted at Shifa ul Mulk Memorial Hospital-Hamdard University and Haidery Herbal Care-North Nazimabad to evaluate its clinical efficacy.

Diabetes management plays a vital role in effectively controlling the disease and minimizing its complications. Lifestyle management plays significant role in managing blood glucose levels in all age and gender segments. Medications are prescribed to regulate blood glucose levels when lifestyle changes alone are insufficient. Regular monitoring of blood sugar levels, along with other important parameters like blood pressure and cholesterol, helps individuals with diabetes to track their progress and make necessary adjustments to their treatment plans.

Dolabi is a time tested formulation of HLWP and it is being used clinically for more than 05 years at Hamdard Matabs all around Pakistan and clinically found satisfactory. The current study is designed in accordance with ICH GCP E6 protocols as approved by WHO and DRAP. It will enable us to present this safer and locally produced combination for the large community suffering with this condition in improving their lives.

ELIGIBILITY:
Inclusion Criteria:

* Subjects having Type II Diabetes Mellitus.
* Subjects having raised FBS above 120 mg/dl and HbA1C level 6.7 or above.
* Subjects over 30 years of age.
* Subjects agree to use study medicine throughout the study.

Exclusion Criteria:

* Subjects suffering from chronic liver diseases and kidney failure.
* Subjects currently taking any hypoglycemic agent(s).
* Subjects suffering from any type of cancer and any other comorbid condition.
* Subjects having history of adverse drug reaction.
* Pregnant and Lactating mother.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-07-04 (Actual); Primary Completion 2025-07-04 (Estimated); Study Completion 2025-10-03 (Estimated)

PRIMARY OUTCOMES:
Blood Sugars | 12 weeks
  Fasting Blood sugars at baseline and the end of treatment will be assess in (mg/dl).
HbA1C (Glycosylated Hemoglobin) | 12 weeks
  Monitoring of HbA1C at baseline and at the end of treatment. the values of HbA1C will be assess in percentage (%).

CONTACTS AND LOCATIONS:
Locations (1):
- Shifa Ul Mulk Memorial Hospital-Hamdard University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No